CLINICAL TRIAL: NCT03447327
Title: Outcome of Single Burr Hole Under Local Anaesthesia in the Management of Chronic Subdural Hematoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hosni Salama, Assistant professor, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB#3893-03-03-2014
Record Dates: First submitted 2018-02-20; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Chronic Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Trephining

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- operated group (Other): patients undergoing surgery for chronic subdural hematoma by single burr hole under local anaesthesia
  Interventions: Procedure: single burr hole

INTERVENTIONS:
Procedure: single burr hole — patients with CSDH operated by single burr hole craniostomy under local anaesthesia

SUMMARY:
Aim of the work: Is to evaluate the prognosis of single burr hole under local anesthesia in management of CSDH according to clinical picture, risk factors, and age.

DETAILED DESCRIPTION:
Patients and methods: We studied 67 consecutive patients with CSDH operated by single burr hole craniostomy under local anaesthesia from Mars, 2014 to February, 2015 in Zagazig University Hospitals according to the aetiology, clinical picture, risk factors, and complications.

ELIGIBILITY:
Inclusion Criteria:chronic subdural hematoma above 19 years old -

Exclusion Criteria:age below 19 years acute subduralhematoma uncoperative patients

-

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-03-05 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2015-08-28 (Actual)

PRIMARY OUTCOMES:
Glasgow Outcome Scale | 6 months postoperative
  The Glasgow Outcome Scale was used as measuremabilityent for neurological oucome after surgery.The patients were classified as as dead, persistant vegetative state, severe disability, moderate disability, and mild dis

IPD SHARING:
Plan to Share IPD: Undecided